CLINICAL TRIAL: NCT02877030
Title: Sensorimotor Exercises in Virtual Reality Platform and Balance in Individuals With Human T-lymphotropic Virus
Brief Title: Sensorimotor Exercises in Virtual Reality Platform in Individuals With Human T-lymphotropic Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pedreira, Érika, M.D. (Individual)
Responsible Party: Principal Investigator, Érika Pedreira, M.D., Pedreira, Érika, M.D.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PedreiraE
Record Dates: First submitted 2016-08-11; First posted 2016-08-24 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2018-05

CONDITIONS: HTLV-1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test control group (Experimental): Start the sensorimotor exercises protocol with video game immediately after the first evaluation
  Interventions: Other: Video game
- Control test group (Active Comparator): Start of sensorimotor exercises with video game protocol after ten weeks
  Interventions: Other: Video game
- comparison group (No Intervention): No intervention

INTERVENTIONS:
Other: Video game — The protocol sensorimotor exercises consist of a virtual game that attaches to the Nintendo Wii and using arrows that are thrown from above, players must perform weight-shifting movements in the Nintendo platform to the target be directed to the trajectory the arrows. The goal is to catch as many arrows.
  Arms: Control test group; Test control group

SUMMARY:
Testing the effectiveness of an exercise protocol engines sensory performed through a virtual reality platform in individuals infected with HTLV-1

DETAILED DESCRIPTION:
Crossover randomized clinical trial to be conducted with people having a previous diagnosis of HTLV-1, they can remain in standing position without assistance. They will be excluded from those presenting amputation of the lower limbs, pregnancy, psychiatric disorders, rheumatic or orthopedic diseases, other neurological disorders associated and those that are experiencing difficulty in understanding the assessment tools used. They will also be recruited to a comparative group, healthy individuals, matched for sex, age and education level. It will be performed three assessments, before randomization, after 10 weeks and after 20 weeks, which will be evaluated in balance, functional mobility, gait and posture. The participants infected with HTLV-1, will be divided into two groups by random distribution, a group will begin the treatment protocol with video game immediately after the first evaluation and the other after ten weeks, with the crossing of the groups . Concealment of allocation will be guaranteed to the examiners who will have no contact with the physiotherapist who will apply the exercise protocol and the team member responsible for drawing. Patients will also be instructed to maintain confidentiality of the entry in the exercise program to other patients and examiners.

ELIGIBILITY:
Inclusion Criteria:

* people having a previous diagnosis of HTLV-1, which can remain in standing position without assistance.

Exclusion Criteria:

* amputation of the lower limbs, pregnancy, psychiatric disorders, rheumatic or orthopedic diseases, other neurological disorders associated and those that are experiencing difficulty in understanding the assessment tools used.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Timed up and Go | average 8 weeks
  Functional mobility in patients with HTLV-1 undergoing rehabilitation with video game
Gait performance at CvMob (Software for movement analysis) | an average 8 weeks
  Gait performance in patients with HTLV-1 undergoing rehabilitation with video game
Posture analysis at CvMob (Software for movement analysis) | average 8 weeks
  Posture analysis in patients with HTLV-1 undergoing rehabilitation with video game

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | average 8 weeks
  Pain in patients with HTLV-1 undergoing rehabilitation with video game
WHOQOL BRIEF | average 8 weeks
  Quality of life in patients with HTLV-1 undergoing rehabilitation with video game

CONTACTS AND LOCATIONS:
Overall Officials: Erika Fonseca, M.D., Principal Investigator — Pedreira, Érika, M.D.
Locations (1):
- Universidade Católica do Salvador, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patricio NA, Vidal DG, Pinto EB, Sa KN, Baptista AF. Effectiveness of virtual reality games for falls, postural oscillations, pain and quality of life of individual HAM/TSP: a randomized, controlled, clinical trial. J Neurovirol. 2020 Oct;26(5):676-686. doi: 10.1007/s13365-020-00880-x. Epub 2020 Jul 31. PMID 32737862